CLINICAL TRIAL: NCT01459224
Title: Whole Body Functional and Anatomical MRI: Accuracy in Staging and Treatment Response Monitoring in Adolescent Hodgkin's Lymphoma Compared to Conventional Multimodality Imaging
Brief Title: MELT - MRI Evaluation of Lymphoma Treatment
Acronym: MELT
Status: Completed | Type: Observational
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: UCL10/0271; CRUK ASC 12707 (Other Grant/Funding Number: Cancer Research UK)
Record Dates: First submitted 2011-10-19; First posted 2011-10-25 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Lymphoma, Hodgkin
MeSH Terms: conditions — Hodgkin Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Patients who are newly diagnosed with Hodgkin's lymphoma will undergo disease staging at diagnosis and initial treatment response assessment. At each time point (initial staging and treatment response assessment) in addition to standard imaging investigations (PET CT, Chest CT, anatomical MRI of the abdomen and pelvis and abdominal USS), patients will undergo an extended MRI scan.

DETAILED DESCRIPTION:
The trial will be a single centre cohort study in patients newly diagnosed with Hodgkin's lymphoma undergoing disease staging at diagnosis and initial treatment response assessment. At each time point (initial staging and treatment response assessment) in addition to standard imaging investigations (PET CT, Chest CT, anatomical MRI of the abdomen and pelvis and abdominal USS), patients will undergo advanced anatomical and functional MRI sequences.

ELIGIBILITY:
Inclusion Criteria:

* Aged 5 to 20 years (inclusive) with participant and parent/guardian informed consent
* Histologically confirmed first presentation of Hodgkin's Lymphoma
* Either entered into the Euronet PHL-C1 trial or LP1 trials OR not formally entered into the Euronet trials but treated on the chemotherapy regimens of the Euronet trials for classical and lymphocyte predominant Hodgkin Lymphoma

Exclusion Criteria:

* Contraindications to MRI (e.g. pacemaker)
* Previous malignancy or previous chemotherapy or radiotherapy treatment for malignancy
* Pregnancy or nursing

Ages: 5 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Hodgkin's Lymphoma
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2011-09; Primary Completion 2014-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
The per site sensitivity and specificity of MRI for both nodal and extranodal sites and concordance in final disease stage with the multi-modality reference standard | The recruited patients to be followed up for 1 year

SECONDARY OUTCOMES:
The number of correct patient classifications into therapy responders and non-responders by MRI compared to the multi modality reference | The recruited patients to be followed up for 1 year
Inter observer agreement for MRI between reporting radiologists (on site and off site). responders by MRI compared to the multi modality reference | The recruited patients to be followed up for 1 year
Sensitivity, specificity of qualitative assessment of Minimum intensity projection (MIP) inverted high B value datasets | The recruited patients to be followed up for 1 year
Utility of apparent diffusion coefficient (ADC) histogram analysis for identifying responsive nodal disease | The recruited patients to be followed up for 1 year
Simulated effect of MRI on clinical management via external oncologic review | The recruited patients to be followed up for 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Stuart A Taylor, Prof, Principal Investigator — UCLH
Locations (1):
- University College London Hospital (UCLH), London, United Kingdom

REFERENCES:
- See also: Coordinating Centre Website — http://www.ctc.ucl.ac.uk/